CLINICAL TRIAL: NCT05148585
Title: Efficacy Of Activity-Based Intervention On Activity, Participation And Kinesiophobia In Patients With Flexor Tendon Injury
Brief Title: Efficacy Of Activity-Based Intervention On Activity, Participation And Kinesiophobia In Patients With Tendon Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sumeyye Cildan Uysal, MSc, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60116787-020/1696
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Flexor Tendon Rupture
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomised-controlled trial group 1 (get only physiotherapy) After flexor tendon repair patients start getting physiotherapy. They use static dorsal splint.
  exercises are progressive according to the healing process. Physiotherapy lasts 12 weeks. then follow-up sixth months.
  group 2 (get both physiotherapy and activity-based therapy) After flexor tendon repair patients start getting physiotherapy. They use static dorsal splint.
  exercises are progressive according to the healing process. Physiotherapy lasts 12 weeks. then follow-up sixth months. Additionally group 2 gets activity-based therapy once a week about an hour. activities are also progressive according to the patients needs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): group 1 (get only physiotherapy) After flexor tendon repair patients start getting physiotherapy. They use static dorsal splint.
  exercises are progressive according to the healing process. Physiotherapy lasts 12 weeks. Then follow-up sixth months.
  Interventions: Other: physiotherapy
- group 2 (Experimental): group 2 (get both physiotherapy and activity-based therapy) After flexor tendon repair patients start getting physiotherapy. They use a static dorsal splint.
  Exercises are progressive according to the healing process. Physiotherapy lasts 12 weeks. then follow-up sixth month. Additionally, group 2 gets activity-based therapy once a week about an hour. activities are also progressive according to the patients needs.
  Interventions: Other: physiotherapy; Other: activity-based therapy

INTERVENTIONS:
Other: physiotherapy — Patients get physiotherapy intervention after the surgery. exercises are progressive. sessions start passive range of motion exercises for 5 weeks while they are using a static dorsal splint. then splints are removed and patients start active range of motion exercises. and exercises progress to blocking, tendon gliding and resistive exercises.
Other: activity-based therapy — patients get from the seventh week to the twelfth week an activity-based therapy. Activities are diverse according to the patient's needs. activities have therapeutic efficacy for improving range of motion, tendon gliding and strength.
  Arms: group 2

SUMMARY:
The aim of our study is to determine the effect of activity-based intervention on the activity, participation levels and kinesiophobia (fear of movement) of the patients by evaluating the person, environment and activity using the Person-Environment-Occupation model (PEO) in the rehabilitation of hand forearm flexor tendon injuries.

DETAILED DESCRIPTION:
Our study will be carried out on housewives who were operated by Pamukkale University Education, Application and Research Center Directorate Orthopedics and Traumatology and Plastic, Reconstructive and Aesthetic Surgery Services due to flexor tendon injury in the forearm or hand.

Patients will be evaluated at the 7th, 12th and 24th weeks post-operatively, before the start of the post-operative physiotherapy program.

The data obtained from the study will be analyzed with the PASW Statistics 18 Release 18.0.0 program. Whether the data fit the normal distribution will be determined using the Shapiro-Wilk test. If parametric conditions are not met, Wilcoxon Signed Rank Test and Friedman Analysis of Variance will be used for intragroup comparisons, and Mann-Whitney U Test will be used for intergroup comparisons. Statistical significance level will be taken as p<0.05.

The physiotherapy program will start the post-operative first week for both group. Activity-based therapy group will have activity exercises that is meaningful for the patients, once a week one hour addition to the physiotherapy.

Patients to be included in groups were randomized in a single block order using Random Allocation Software 1.0.0.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-65
* flexor tendon injury
* Primary tendon repair performed
* a woman

Exclusion Criteria:

* Presence of major nerve injury (radial, ulnar, median nerve)
* Presence of concomitant injuries (fracture, joint injury, ligament injury)
* Presence of any previous or ongoing orthopedic, neurological, rheumatological and metabolic disease or disorder in the relevant extremity

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The Canadian occupational performance measure | six month
  The Canadian occupational performance measure, was used to determine the effect of the intervention on the participant's self-determined occupational performance goals. A scale of one to ten was used, where ten was the most important goal needed to be attained by the participants.
  Using the same scale, the participants were asked to rate the performance of the occupations and satisfaction with their performance. Both the sum of performance and satisfaction scores were divided by the number of identified problems to compute the overall score for analysis.
Tampa Kinesiophobia Scale | six month
  It is a 17-item scale developed to measure fear of movement and/or (re) injury. A high score indicates a high level of kinesiophobia. A score of <37 indicates low kinesiophobia, and a score≥37 indicates a high level of kinesiophobia.

SECONDARY OUTCOMES:
jebsen taylor hand function test | six month
  Jebsen Taylor Hand Function Test: It has 7 subtasks: writing, turning cards, collecting small objects, eating, placing chips, moving empty and full boxes. The test will begin with the non-dominant hand and both hands will be evaluated.
Michigan Hand Outcome Questionnaire: | six month
  It is a hand injury-specific questionnaire developed to measure outcomes for patients with all types of hand disorders.It is a self-filled questionnaire consisting of 6 sections and 57 questions. Scoring ranges from 0-100, with a higher score indicating better condition excluding pain.
grip strength | 6 month
  Pinch Grip Strength: It will be made with three different measurements. Grip strength, Pinch grip, Lateral grip, Triple grip strength: measurements will be made by squeezing the pinch meter between the palmar surface of the thumb, index and middle fingers.
  3 repetitions will be done and the average will be recorded. A one-minute rest period will be given between repetitions.
range of motion | six month
  Metacarpophalangeal, proximal interphalangeal, distal interphalangeal joint flexion-extension, wrist flexion-extension, radial-ulnar deviation movements of the affected finger and finger in the intact extremity will be evaluated with a goniometer.
  Buck Gramcko will be used to score joint range of motion. Makes a score using the pulp-palm distance, combined flexion and extension deficit. There are 2 different scoring systems to be used separately for long fingers and thumb. Classification according to scores; 14-15 points perfect 11-13 points good 7-10 points satisfactory 0-6 points bad
Visual Analog Scale | 7 weeks
  Visual Analog Scale (VAS): "0" denotes when there is no pain, and "10" denotes the most severe pain level perceived. Patients will be asked to mark the intensity of pain they feel during activity, rest and at night on a 10 cm vertical line, and then the pain intensity will be determined by measuring the distance on the line.

CONTACTS AND LOCATIONS:
Overall Officials: Sumeyye CILDAN UYSAL, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only measurements can be shared after the recruitment is finished.
Supporting Information: Study Protocol, SAP
Time Frame: after the study has completed.
Access Criteria: investigation

REFERENCES:
- [Background] Colaianni D, Provident I. The benefits of and challenges to the use of occupation in hand therapy. Occup Ther Health Care. 2010 Apr;24(2):130-46. doi: 10.3109/07380570903349378. PMID 23898899
- [Background] Guzelkucuk U, Duman I, Taskaynatan MA, Dincer K. Comparison of therapeutic activities with therapeutic exercises in the rehabilitation of young adult patients with hand injuries. J Hand Surg Am. 2007 Nov;32(9):1429-35. doi: 10.1016/j.jhsa.2007.08.008. PMID 17996780